CLINICAL TRIAL: NCT05854095
Title: The Study for Evaluation of Acute Phase Safety and Efficacy of 'Pivot Bridge' to Short-term Treat Functional Tricuspid Regurgitation : Multi-center, Open Label, Single Arm, Investigator Initiated Exploratory Pilot Study
Brief Title: The Study for Evaluation of Acute Phase Safety and Efficacy of 'Pivot Bridge' to Short-term Treat FTR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tau-MEDICAL Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Joo Yong Hahn, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pivot Bridge-FIM
Record Dates: First submitted 2023-01-30; First posted 2023-05-11 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Functional Tricuspid Regurgitation
Keywords: FTR; RV failure; TauPnu

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pivot Bridge (Experimental): transcatheter for short-term treat Functional Tricuspid regurgitation
  Interventions: Device: Pivot Bridge

INTERVENTIONS:
Device: Pivot Bridge — transcatheter for short-term treat Functional Tricuspid regurgitation

SUMMARY:
evaluation of safety and efficacy of 'Pivot Bridge' to short-term treat Functional Tricuspid regurgitation

DETAILED DESCRIPTION:
evaluation of safety and efficacy of 'Pivot Bridge' to short-term treat Functional Tri cuspid regurgitation : multi-center, open label, single arm, investigator initiated exploratory pilo t study

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females aged 20 years or above
* Patients with clinical symptoms (Symptomatic) whose degree of tricuspid regurgitation using echocardiography meets the criteria of Severe or higher presented in the TR grade classification table
* Short-term treatment using a catheter is required (expected to be effective) by a local site heart team including at least one cardiothoracic (cardiovascular) specialist and at least one thoracic surgeon each, and clinical symptoms of NYHA Class Ⅱ or higher person who falls under
* In the screening test, A person who can confirm the possibility of reducing tricuspid valve regurgitation by inserting that 'Pivot Balloon' (Clinical Trial Approval No. 1327), etc.) through the same access path as the 'Pivot Bridge', a clinical trial medical device
* An individual who voluntarily agreed to the participation in the clinical trial and signed the written consent
* An individual who is able to understand and comply with the instructions and who can participate in the period before the clinical trial

Exclusion Criteria:

* Uncontrolled hyperthyroidism
* A recent formation of soft blood clot or embolic material
* Uncorrected coagulopathy
* Prohibition of anticoagulant agents
* Those who had experience with anticoagulant use prior to participation in this clinical trial and who were treated with major bleeding (minor bleeding such as nosebleeds that can be hemostasis not applicable) due to anticoagulant use at this time or accompanied by severe anemia requiring hospitalization one with experience
* Previous insertion of a device such as an Implantable Cardioverter Defibrillator (ICD) or a pacemaker
* Those who is judged to have little possibility of reducing tricuspid valve regurgitation by inserting a balloon-type device (e.g. ASD sizing balloon, pivot balloon, etc.) through the same access route as the clinical trial medical device 'Pivot Bridge'
* Persons with an anatomical structure that cannot be inserted through the corresponding route

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2023-12-27 (Actual)

PRIMARY OUTCOMES:
Assessment of Acute phase safety | immediately after the procedure
  Check all adverse reactions Including serious adverse events and serious adverse medical device reactions

SECONDARY OUTCOMES:
Efficacy endpoint-1: Changes of hemodynamics | within 1week of implant
  Echocardiogram: Pulmonay artery forward flow(RV stroke volume) in ml
Efficacy endpoint-1: Changes of hemodynamics(1) | within 1week of implant
  Echocardiogram: RV Cardiac output(Heart rate x RVOT area x RVOT TVI) in ml/min
Efficacy endpoint-1: Changes of hemodynamics(2) | within 1week of implant
  Echocardiogram: Fractional area change in percentage
Efficacy endpoint-1: Changes of hemodynamics(3) | within 1week of implant
  Echocardiogram: LVEF in percentage
Efficacy endpoint-1: Changes of hemodynamics(4) | within 1week of implant
  Echocardiogram: Peak systolic annular velocity in cm/sec
Efficacy endpoint-1: Changes of hemodynamics(5) | within 1week of implant
  Echocardiogram: Tricuspid annular plane systolic excursion(TAPSE) in mm
Efficacy endpoint-1: Changes of hemodynamics(6) | within 1week of implant
  Echocardiogram: LVOT stroke volume in ml
Efficacy endpoint-1: Changes of hemodynamics(7) | within 1week of implant
  Echocardiogram: TV annular diameter in mm
Efficacy endpoint-1: Changes of hemodynamics(8) | within 1week of implant
  Echocardiogram: RV diameter base in mm
Efficacy endpoint-1: Changes of hemodynamics(9) | within 1week of implant
  Echocardiogram: Inferior vena cava diameter and PW tracing - Assessment of the presence or absence of systolic flow reversal
Efficacy endpoint-1: Changes of hemodynamics(10) | within 1week of implant
  Echocardiogram: RV-RA coupling(Tapse/PASP) in ratio
Efficacy endpoint-1: Changes of hemodynamics(11) | within 1week of implant
  Cardiac CT : RV volume in ml
Efficacy endpoint-2: Technical feasibility and TR grade changes | within 1week of implant
  Evaluation of reduction in tricuspid regurgitation grade (TR grade) according to Echo parameters
Assessment of short-term safety | within 1week of implant
  Check all adverse reactions Including serious adverse events and serious adverse medical device reactions

CONTACTS AND LOCATIONS:
Overall Officials: Joo-Yong Hahn, PhD, Principal Investigator — Samsung Medical Center
Locations (10):
- South Korea (10):
  - Keimyung University Dongsan Hospital, Daegu, Dalseo-gu
  - Hallym University Medical Center, Anyang, Dongan-gu
  - Soonchunhyang University Bucheon Hospital, Bucheon-si, Gyeonggi-do
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Chungnam National University Hospital (CNU Hospital), Daejeon, Jung-gu
  - Chungnam National University sejong Hospital, Daejeon, Jung-gu
  - Ulsan Hospital, Ulsan, Nam-gu
  - Asan Medical Center, Seoul, Songpa-gu
  - Bucheon Sejong Hospital, Bucheon-si
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chaabane C, Otsuka F, Virmani R, Bochaton-Piallat ML. Biological responses in stented arteries. Cardiovasc Res. 2013 Jul 15;99(2):353-63. doi: 10.1093/cvr/cvt115. Epub 2013 May 10. PMID 23667187
- [Background] Hwang HY, Kim KH, Kim KB, Ahn H. Treatment for severe functional tricuspid regurgitation: annuloplasty versus valve replacement. Eur J Cardiothorac Surg. 2014 Aug;46(2):e21-7. doi: 10.1093/ejcts/ezu224. Epub 2014 Jun 10. PMID 24917649
- [Background] Groves PH, Lewis NP, Ikram S, Maire R, Hall RJ. Reduced exercise capacity in patients with tricuspid regurgitation after successful mitral valve replacement for rheumatic mitral valve disease. Br Heart J. 1991 Oct;66(4):295-301. doi: 10.1136/hrt.66.4.295. PMID 1747281
- [Background] Rommel KP, Besler C, Noack T, Blazek S, von Roeder M, Fengler K, Ender J, Gutberlet M, Desch S, Borger MA, Thiele H, Lurz P. Physiological and Clinical Consequences of Right Ventricular Volume Overload Reduction After Transcatheter Treatment for Tricuspid Regurgitation. JACC Cardiovasc Interv. 2019 Aug 12;12(15):1423-1434. doi: 10.1016/j.jcin.2019.02.042. Epub 2019 Jul 17. PMID 31326430
- [Background] Kelly BJ, Ho Luxford JM, Butler CG, Huang CC, Wilusz K, Ejiofor JI, Rawn JD, Fox JA, Shernan SK, Muehlschlegel JD. Severity of tricuspid regurgitation is associated with long-term mortality. J Thorac Cardiovasc Surg. 2018 Mar;155(3):1032-1038.e2. doi: 10.1016/j.jtcvs.2017.09.141. Epub 2017 Nov 8. PMID 29246545
- [Background] Taramasso M, Benfari G, van der Bijl P, Alessandrini H, Attinger-Toller A, Biasco L, Lurz P, Braun D, Brochet E, Connelly KA, de Bruijn S, Denti P, Deuschl F, Estevez-Loureiro R, Fam N, Frerker C, Gavazzoni M, Hausleiter J, Ho E, Juliard JM, Kaple R, Besler C, Kodali S, Kreidel F, Kuck KH, Latib A, Lauten A, Monivas V, Mehr M, Muntane-Carol G, Nazif T, Nickening G, Pedrazzini G, Philippon F, Pozzoli A, Praz F, Puri R, Rodes-Cabau J, Schafer U, Schofer J, Sievert H, Tang GHL, Thiele H, Topilsky Y, Rommel KP, Delgado V, Vahanian A, Von Bardeleben RS, Webb JG, Weber M, Windecker S, Winkel M, Zuber M, Leon MB, Hahn RT, Bax JJ, Enriquez-Sarano M, Maisano F. Transcatheter Versus Medical Treatment of Patients With Symptomatic Severe Tricuspid Regurgitation. J Am Coll Cardiol. 2019 Dec 17;74(24):2998-3008. doi: 10.1016/j.jacc.2019.09.028. Epub 2019 Sep 27. PMID 31568868
- [Background] Kolte D, Elmariah S. Current state of transcatheter tricuspid valve repair. Cardiovasc Diagn Ther. 2020 Feb;10(1):89-97. doi: 10.21037/cdt.2019.09.11. PMID 32175231
- [Background] Izumi C. Isolated functional tricuspid regurgitation: When should we go to surgical treatment? J Cardiol. 2020 Apr;75(4):339-343. doi: 10.1016/j.jjcc.2019.11.001. Epub 2019 Nov 29. PMID 31787551
- [Background] Henning RJ. Tricuspid valve regurgitation: current diagnosis and treatment. Am J Cardiovasc Dis. 2022 Feb 15;12(1):1-18. eCollection 2022. PMID 35291509
- [Background] Asmarats L, Puri R, Latib A, Navia JL, Rodes-Cabau J. Transcatheter Tricuspid Valve Interventions: Landscape, Challenges, and Future Directions. J Am Coll Cardiol. 2018 Jun 26;71(25):2935-2956. doi: 10.1016/j.jacc.2018.04.031. PMID 29929618
- [Background] Taramasso M, Hahn RT, Alessandrini H, Latib A, Attinger-Toller A, Braun D, Brochet E, Connelly KA, Denti P, Deuschl F, Englmaier A, Fam N, Frerker C, Hausleiter J, Juliard JM, Kaple R, Kreidel F, Kuck KH, Kuwata S, Ancona M, Malasa M, Nazif T, Nickenig G, Nietlispach F, Pozzoli A, Schafer U, Schofer J, Schueler R, Tang G, Vahanian A, Webb JG, Yzeiraj E, Maisano F, Leon MB. The International Multicenter TriValve Registry: Which Patients Are Undergoing Transcatheter Tricuspid Repair? JACC Cardiovasc Interv. 2017 Oct 9;10(19):1982-1990. doi: 10.1016/j.jcin.2017.08.011. PMID 28982563
- [Background] Curio J, Demir OM, Pagnesi M, Mangieri A, Giannini F, Weisz G, Latib A. Update on the Current Landscape of Transcatheter Options for Tricuspid Regurgitation Treatment. Interv Cardiol. 2019 May 21;14(2):54-61. doi: 10.15420/icr.2019.5.1. eCollection 2019 May. PMID 31178930
- [Background] Park SJ, Oh JK, Kim SO, Lee SA, Kim HJ, Lee S, Jung SH, Song JM, Choo SJ, Kang DH, Chung CH, Song JK, Lee JW, Kim DH, Kim JB. Determinants of clinical outcomes of surgery for isolated severe tricuspid regurgitation. Heart. 2021 Mar;107(5):403-410. doi: 10.1136/heartjnl-2020-317715. Epub 2020 Nov 2. PMID 33139325
- [Background] Hahn RT, Meduri CU, Davidson CJ, Lim S, Nazif TM, Ricciardi MJ, Rajagopal V, Ailawadi G, Vannan MA, Thomas JD, Fowler D, Rich S, Martin R, Ong G, Groothuis A, Kodali S. Early Feasibility Study of a Transcatheter Tricuspid Valve Annuloplasty: SCOUT Trial 30-Day Results. J Am Coll Cardiol. 2017 Apr 11;69(14):1795-1806. doi: 10.1016/j.jacc.2017.01.054. PMID 28385308